CLINICAL TRIAL: NCT03770143
Title: Evaluation of the Effect of Palm Olein Free Formula on Intestinal Flora and Gastrointestinal Tolerance
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Merih Cetinkaya, Associate Professor, MD,PhD, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: ANCL034
Record Dates: First submitted 2016-05-11; First posted 2018-12-10 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2018-12

CONDITIONS: Feeding; Disorder, Nonorganic Origin; Calcium Disorder; Intestinal Bacteria Flora Disturbance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Group 1: Infants feeding predominantly with palm olein free formula if presence in addition to breast milk for 8 weeks of life
  Interventions: Other: Feeding with palm olein formula
- Group 2: Infants feeding with other formulas including palm olein if presence in addition to breast milk for 8 weeks of life
- Group 3: Having similar demographical properties with infants feeding with breast milk (gender, age, weight, height)

INTERVENTIONS:
Other: Feeding with palm olein formula
  Groups: Group 1

SUMMARY:
Depending on recent studies in literature the investigators aimed to compare whether gastrointestinal tolerance differs between infants fed with palm olein containing or palm olein free formulas. Besides it is showed that palm olein containing formulas decreases the absorption of fat and calcium by forming insoluble calcium soaps. So it is suggested that intestinal flora might be affected as a reason of these specialties. This study also aimed to investigate with culture-independent methods whether feeding infants with palm olein free formula results in the modification of their intestinal microbiota in such a way that is similar to breastfed ones.

DETAILED DESCRIPTION:
Recent studies in literature the investigators aimed to compare whether gastrointestinal tolerance differs between infants fed with palm olein containing or palm olein free formulas. Besides it is showed that palm olein containing formulas decreases the absorption of fat and calcium by forming insoluble calcium soaps. So it is suggested that intestinal flora might be affected as a reason of these specialties. This study also aimed to investigate with culture-independent methods whether feeding infants with palm olein free formula results in the modification of their intestinal microbiota in such a way that is similar to breastfed ones.

ELIGIBILITY:
Inclusion Criteria:

The data of the patients who fulfilled the following criteria are evaluated.

1. Term infants between 38 and 40 weeks of gestational age and/or with a birth weight of > 2500grams who are either breastfed or formula fed.

   Selection of the subgroup using oral nutrition
2. Feeding predominantly with palm olein free formula if presence in addition to breast milk for 8 weeks of life
3. Feeding with other formulas including palm olein if presence in addition to breast milk for 8 weeks of life Selection of the subgroup not using oral nutritional supplement (control group)
4. Having similar demographical properties with infants feeding with breast milk (gender, age, weight, height)

Exclusion Criteria:

* Infants with major congenital abnormalities will be excluded.
* Infants with lack of data will also be excluded.
* Infants, whose parents don't agree with informed consent, will be excluded.

Max Age: 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: A total of 90 healthy infants (30 under breast-feeding, 30 feeding with palm olein free formula and 30 feeding with palm olein formula) will be included. Infants feeding enterally more than %70 with breast milk will be considered as breast-feeding. Infants who had not adequate weight gain and need formula will be randomized to receive either palm olein or palm olein free term formula in addition to mother milk. Parental informed consent will be taken and infants whose parents give permission will be included.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2016-05; Primary Completion 2016-08 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Stool consistency | 10 weeks
  Amsterdam Infant Stool Scale

SECONDARY OUTCOMES:
Bacteria Count | 10 weeks
  number of the copy of DNA of Intestinal Flora Content

CONTACTS AND LOCATIONS:
Overall Officials: Seda Yilmaz Semerci, Study Director — Kanuni SSTRH
Locations (1):
- Kanuni Sultan Suleyman Training and Research Hospital, Istanbul, Kucukcekmece, Turkey (Türkiye)